CLINICAL TRIAL: NCT04644627
Title: TOPICAL GENTAMICIN TREATMENT OF PATIENTS WITH EPIDERMOLYSIS BULLOSA DUE TO NONSENSE MUTATIONS
Brief Title: Topical Gentamicin Nonsense Suppression Therapy of EB
Acronym: GENTELBULL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Øystein Sandanger, Principal Investigator, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105989
Record Dates: First submitted 2020-11-20; First posted 2020-11-25 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa | interventions — Gentamicins

STUDY DESIGN:
Intervention Model Description: Each patient serve as its own control, study treatment is given to one half of the body, the other half receives regular wound treatment. Which side to be treated is determined with randomization.
Masking Description: Wound size calculations will be performed on digital photos, the outcome assessor will not know which wounds are treated and which are controls.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Each patient serves as its own control: one half is treated with the study treatment in addition to standard wound therapy, the other half receives standard wound therapy only.
  Interventions: Drug: Gentamicin Sulfate

INTERVENTIONS:
Drug: Gentamicin Sulfate — Topical gentamicin ointment on wounds once daily for 6 weeks

SUMMARY:
The overall purpose of this study is to address whether topical gentamicin therapy is an effective and feasible treatment. Specifically, we will investigate the effect of non-intensive treatment (once daily or every other day) on skin protein expression, as well as quantify the effect on wound healing in patients with EB caused by PSC (part A). Furthermore, we will address in vitro whether gentamicin restores protein expression of genes affected by SSM in fibroblasts derived from skin biopsies obtained from patients with EB caused by SSM (part B). If these in vitro experiments yield positive results, the patients donating the cells will be offered to enter part A of this study. The overall duration of part A in this study is planned to be 18 weeks per patients and consists of a 6 weeks treatment period followed by a 12 week follow up period. Each patient will attend 3 study visits: at week 0, week 6 and week 18. All patients will be included within a time period of 12 months. The overall duration of part B will be up to 8 weeks per patients of which 4-7 weeks are spent to prepare fibroblasts obtained from skin biopsies. Then 5 days of in vitro intervention and subsequent analysis follows. Altogether, the duration of the GENTELBULL study will be 78 weeks or less.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has EB caused by nonsense mutation
2. The patient has a symmetrical distribution of wounds which allows for wounds on one side of the body to serve as control wounds, while study therapy is applied to the other side.
3. The patient (if an adult) or parent(s)/guardian(s) is capable of giving signed informed consent as described in Appendix 1 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
4. Women of childbearing potential must use a highly effective contraception method

Exclusion Criteria:

1. Known contact allergy against gentamicin sulfate or other ingredients in the ointment
2. Known intolerance to gentamicin sulfate of any sort
3. Moderate or severely reduced kidney function (eGFR <45)
4. Use other experimental therapy against EB
5. Receiving systemic aminoglycosides during the last 3 months
6. The patient uses muscle relaxant drug(s)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Wound size reduction | 6 weeks
  Mean of ratios for wound areas (measured in cm2) at week 6 to that of week 0 of gentamicin-treated wounds, compared to the corresponding mean of ratios for standard care-treated wounds. The observed effect is considered significant if p<0.05 (unpaired t-test). Of note, each patient may or may not reach the primary end point independent of the other participants

SECONDARY OUTCOMES:
Healed skin robustness | 18 weeks
  Mean of ratios for single wound areas (measured in cm2) at week 18 to that of week 6 of gentamicin-treated wounds, compared to the corresponding mean of ratios for standard care-treated wounds. The observed effect is considered significant if p<0.05 (unpaired t-test). Of note, each patient may or may not reach the primary end point independent of the other participants
Systemic gentamicin levels | 6 weeks
  Trough levels gentamicin in serum day 1 and week 6. If detectable day 1, levels will be monitored more frequently
Protein restoration by gentamicin | 6 weeks
  Immune histochemistry analysis of skin biopsy obtained from healed treated wound area at week 6 and 18 compared to skin biopsy from non-treated non-affected skin obtained at baseline (negative control) and non-affected skin from one healthy control (positive control)

CONTACTS AND LOCATIONS:
Overall Officials: Øystein Sandanger, MD, PhD, Principal Investigator — Section of Dermatology, OUS
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No